CLINICAL TRIAL: NCT00022607
Title: Phase II Randomized Trial of Bevacizumab Versus Bevacizumab and Thalidomide for Relapsed/Refractory Multiple Myeloma
Brief Title: Bevacizumab With or Without Thalidomide in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: California Cancer Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068834; CCC-PHII-30; CHNMC-PHII-30; CHNMC-IRB-01006; NCI-2712
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2004-10

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bevacizumab; Thalidomide

INTERVENTIONS:
Biological: bevacizumab
Drug: thalidomide

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. Thalidomide may stop the growth of cancer cells by stopping blood flow to the tumor. It is not yet known whether bevacizumab works better with or without thalidomide for multiple myeloma.

PURPOSE: This randomized phase II trial is to see if bevacizumab works better with or without thalidomide in treating patients who have relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response rate and time to progression in patients with relapsed or refractory multiple myeloma treated with bevacizumab with or without thalidomide.
* Compare the toxicity of these regimens in these patients.
* Compare the effects of these regimens on histological and molecular biomarkers of angiogenesis, tumor invasion, and cell death in these patients.
* Correlate plasma and urine vascular endothelial growth factor and basic fibroblast growth factor levels and other potential markers of angiogenesis and myeloma cell proliferation with outcome in patients treated with these regimens.
* Determine the pharmacokinetics of thalidomide in these patients.
* Compare the effects of these regimens on the psychological/physical well being of these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior treatment with thalidomide (yes vs no).

Patients who have received no prior treatment with thalidomide are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive bevacizumab IV over 30-90 minutes on days 1, 15, 29, and 43. Patients also receive oral thalidomide once daily.
* Arm II: Patients receive bevacizumab as in arm I. Patients who have received prior treatment with thalidomide receive bevacizumab as in arm I.

Courses repeat every 56 days in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly for 3 months and then every 3-4 months for 3 years.

PROJECTED ACCRUAL: A total of 55-103 patients (16-32 who have received prior thalidomide, 16-32 in arm I, and 23-39 in arm II) will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed progressing multiple myeloma

  * Stages I, II, or III
  * More than 25% increase in urine or plasma paraprotein levels
  * More than 5% malignant plasma cell involvement in bone marrow
* Smoldering myeloma is eligible provided there is evidence of progressive disease requiring therapy

  * At least 25% increase in M protein levels or Bence Jones excretion
  * Hemoglobin no greater than 10.5 g/dL
  * Frequent infections
  * Hypercalcemia
  * Rise in serum creatinine above normal on 2 separate occasions
* Nonsecretory multiple myeloma that is bidimensionally measurable by MRI or CT scan is eligible provided the disease site is new or has shown an increase in M protein levels or Bence Jones excretion is greater than 30% from baseline
* No prior or concurrent CNS involvement with primary or metastatic tumor
* No nonquantifiable monoclonal proteins or IgM peaks unless there is evidence of bidimensionally measurable disease by MRI or CT scan
* No history of hemorrhagic tumor or hemorrhagic metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* See Disease Characteristics
* Absolute neutrophil count ≥1,000/mm^3
* Platelet count ≥ 50,000/mm^3
* No hemorrhagic illness within the past 3 weeks

Hepatic:

* Bilirubin ≤ 1.5 mg/dL
* SGOT/SGPT≤ 2.5 times upper limit of normal (ULN)
* INR ≤ 1.5
* aPTT < 1.5 times ULN

Renal:

* See Disease Characteristics
* Creatinine ≤ 2 mg/dL
* Creatinine clearance ≥ 40 mL/min
* Calcium ≤ 12 mg/dL
* No nephrotic syndrome

Cardiovascular:

* No active coronary artery disease
* No New York Heart Association class II-IV congestive heart failure
* No grade II or greater peripheral vascular disease (i.e, ischemic rest pain, non-healing ulcer, or tissue loss)
* No uncontrolled hypertension
* No history of deep venous thrombosis
* No vascular illness within the past 3 weeks
* No arterial thromboembolic event within the past 6 months, including any of the following:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina
  * Myocardial infarction

Pulmonary:

* No history of pulmonary embolus

Other:

* No other prior malignancy unless the patient has been in complete remission for at least 2 years
* No peripheral neuropathy or CNS abnormalities ≥ grade 2

  * Patients with prior exposure to thalidomide and assigned to arm I may have grade 2 peripheral or CNS abnormalities
* No seizure disorder
* No serious non-healing wound, ulcer, or bone fracture
* No trauma within the past 3 weeks
* No significant inflammatory illness within the past 3 weeks
* No known hypersensitivity to Chinese hamster ovary cell products
* No known hypersensitivity to other recombinant human or humanized antibodies and/or positive human antimurine antibodies/human antichimeric antibodies
* No other significant medical, psychological, or social problem that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for at least 2 weeks before and during study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Chemotherapy
* Prior nonmyeloablative transplantation allowed provided the following are true:

  * Patient is not receiving concurrent immunosuppressive therapy
  * Patient has no signs of graft-versus-host disease
* Concurrent epoetin alfa allowed if started at least 4 weeks prior to study entry

Chemotherapy:

* No more than 5 prior chemotherapy regimens

  * Thalidomide, steroids, and interferon are not considered part of prior regimens
  * Mobilization with chemotherapy followed by either single or tandem autologous transplantation is counted as 1 prior regimen
  * Mobilization with chemotherapy followed by autologous and subsequent nonmyeloablative HLA-matched sibling allogeneic transplantation is counted as 1 prior regimen
* At least 3 weeks since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* See Chemotherapy
* At least 2 weeks since prior steroids
* No concurrent steroids

Radiotherapy:

* At least 3 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* At least 3 weeks since prior surgery, including biopsy of a visceral organ

Other:

* At least 10 days since prior anticoagulants, including aspirin
* At least 2 days since prior nonsteroidal anti-inflammatory agents
* Concurrent bisphosphonates allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01; Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - University of Chicago Cancer Research Center, Chicago, Illinois